CLINICAL TRIAL: NCT03888274
Title: ClearUP Longitudinal Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tivic Health Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP00003
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Sinus Pain; Congestion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active (Experimental)
  Interventions: Device: ClearUP Sinus Pain Relief

INTERVENTIONS:
Device: ClearUP Sinus Pain Relief — Microcurrent Device Treatment

SUMMARY:
Single arm, open label pilot study assessing the longitudinal home use of ClearUp Sinus Pain Relief for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-71 years of age (inclusive)
* Present with symptoms of sinus pain or facial pain in the forehead, periorbital, facial, or nasal region
* Current pain score ≥ 5 (Numeric Rating Scale 0-10)
* Frequency of sinus/facial pain at least twice weekly for 1 month
* Able to read and understand English
* Agree to participate in the study
* Able and willing to provide Informed Consent

Exclusion Criteria:

* Do not meet Inclusion Criteria
* Currently taking or recently taken any oral steroid medications in the last 90 days
* Sinus surgery in previous 90 days
* History of Chronic Migraine (≥ 15 headache days per month)
* Pain location in the vertex, occiput, or temporal region of the skull or in mandibular region
* Purulent rhinorrhea

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy and Asthma Associates of Santa Clara Valley Research Center, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldsobel AB, Prabhakar N, Gurfein BT. Prospective trial examining safety and efficacy of microcurrent stimulation for the treatment of sinus pain and congestion. Bioelectron Med. 2019 Nov 20;5:18. doi: 10.1186/s42234-019-0035-x. eCollection 2019. PMID 32232107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale for Pain
Description: Change in Numeric Rating Scale for Pain from Baseline to Four Weeks. Scale range 0, no pain, to 10 severe pain.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 30
score on a scale
  Baseline | 6.5 (0.20)
  4 Weeks | 3.6 (0.36)

2. Secondary Outcome: Congestion Quantifier 7
Description: Change in Congestion Quantifier 7 from Baseline to Four Weeks. Congestion Quantifier 7 is a 7 item questionnaire that quantifies congestion symptom severity. It is scored from 0 (no congestion symptoms) to 28 (severe congestions symptoms).
Time Frame: 4 Weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 30
score on a scale
  Baseline | 18.1 (0.85)
  4 Weeks | 11.0 (1.05)

3. Secondary Outcome: Numeric Rating Scale for Pain
Description: Acute Change in Numeric Rating Scale for Pain from Baseline to 6 Hours. Scale range 0, no pain, to 10 severe pain.
Time Frame: 6 hours
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 30
score on a scale
  Baseline | 6.5 (0.20)
  6 Hours | 4.3 (0.37)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 4 week duration of the study.
Description: A serious adverse event is defined as one that results in death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=30)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 (2) — Mild skin erythema
Headache (Nervous system disorders) | 1 (1)
Eyelid Twitch (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03888274/Prot_SAP_000.pdf